CLINICAL TRIAL: NCT07179172
Title: Neurobiological Investigations of Mindfulness, Depression and Sleep Disturbances in Medical Staffs and Community Elders
Acronym: NIMDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202502057
Record Dates: First submitted 2025-08-24; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Sleep Disturbances; Depression
Keywords: Medical personnel; sleep; depression; mental health; preventive medicine; mindfulness; aging; functional magnetic resonance imaging (fMRI); wearable device
MeSH Terms: conditions — Parasomnias; Depression; Psychological Well-Being | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MBSR group (Experimental): Mindfulness-Based Stress Reduction (MBSR) 8-Week Program
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR) 8-Week Program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) 8-Week Program — The program consists of weekly 2.5-hour sessions over an eight-week period. The certified mindfulness instructor will follow a curriculum that includes in-class formal practice (2.5 hours) and assigned informal practice (30-40 minutes daily).
  During the sessions, the instructor will guide participants through mindfulness meditation, pain awareness, mindful yoga, gratitude practice, loving-kindness meditation, and the sharing of daily life experiences. Additionally, a full-day, eight-hour silent retreat (9 a.m. to 5 p.m.) will be held between weeks six and seven to deepen inner awareness.
  Following each weekly group session, participants will be instructed to perform and self-record daily home practice, which will be discussed and evaluated during the following week's class. The total course duration is approximately 26 hours, and participants will receive a certificate of completion upon graduation.

SUMMARY:
The research team proposes a multi-year study with the first year focusing on the developmental phase. In this initial phase, we aim to recruit 40 participants (including healthcare staff and older adults) from Shuang-Ho Hospital and the surrounding community to undergo two mindfulness intervention sessions, each lasting four months. We anticipate that these interventions will prevent and alleviate stress and depressive symptoms while enhancing self-awareness and psychological health.

DETAILED DESCRIPTION:
Mindfulness-based interventions (MBI) have capability to effectively reduce anxiety, alleviate stress responses, and decrease negative emotional states and rumination. However, the majority of studies have predominantly focused on younger populations or university students, utilizing subjective scales as assessment tools. Noticeable scarcity of studies is in need to implement mindfulness programs among healthcare staff and elderly patients experiencing depression, despite these groups exhibiting urgent needs for improving mental health. This research project aims to introduce MBI within a healthcare setting to effectively alleviate workplace stress, enhance self-awareness, and improve sleep quality or psychological well-being among medical personnel. Additionally, this initiative targets mental health issues in older adults by recruiting participants from the community surrounding Shuang-Ho Hospital. The program aims to prevent depression, delay cognitive decline, and reduce suicide risk while providing continuous opportunities for personal growth among the senior adults. This effort aligns well with Taiwan government initiatives promoting social support and long-term care in the over-aging societies and lays the groundwork for quantitative research on MBI for older adults.

The research team proposes a multi-year study with the first year focusing on the developmental phase. In this initial phase, we aim to recruit 40 participants (including healthcare staff and older adults) from Shuang-Ho Hospital and the surrounding community to undergo two mindfulness intervention sessions, each lasting four months. We anticipate that these interventions will prevent and alleviate stress and depressive symptoms while enhancing self-awareness and psychological health. To explore the neurophysiological effects of mindfulness courses, we will employ advanced technologies, including non-invasive fiber optic physiological monitoring (nFOPT), wearable Garmin smartwatches, and functional magnetic resonance imaging (fMRI), to observe changes in participants' central and peripheral nervous systems throughout the intervention. fMRI will elucidate the central modulatory effects of mindfulness on neural function, while Garmin smartwatches will provide continuous physiological data monitoring. Coupling these methods with nFOPT and the Belun ring will allow for comprehensive sleep quality assessments. This interdisciplinary approach addresses the limitations of prior qualitative-focused mindfulness research. Ultimately, this study aims to advance the care of healthcare workers, fulfill social responsibilities associated with university outreach, and make significant contributions world-wide to both the academic fields of mindfulness and neuroscience.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital staff aged 20-65 years, or elderly individuals aged 55-90 years.
2. Individuals willing to participate in the entire mindfulness course and comply with study enrollment procedures.-

Exclusion Criteria:

1. History of major neurological disorders (e.g., epilepsy, Parkinson's disease, stroke).
2. History of major psychiatric disorders (e.g., schizophrenia, bipolar disorder).
3. Use of medications that may affect sleep, other than illegal substances or sleeping pills.
4. Individuals with metal implants.
5. Individuals with claustrophobia.
6. Pregnant women.
7. History of alcohol or substance addiction.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Taiwan Geriatric depression scale (TGDS) | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  A self-report scale collected through an online questionnaire, with a minimum score of 0 and a maximum score of 15, where higher scores indicate more depressive symptoms.
Pittsburgh Sleep Quality Index (PSQI) | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  A self-report questionnaire that assesses sleep quality and disturbances over a 1-month period. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A global PSQI score greater than 5 suggests poor sleep quality.
The World Health Organization-Five Well-Being Index (WHO-5) | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  A short self-report questionnaire consisting of 5 items that assess subjective psychological well-being over the past two weeks. Each item is scored on a 6-point Likert scale (0 = at no time to 5 = all of the time). The raw total score ranges from 0 to 25, with higher scores indicating better well-being. A score below 13 suggests poor well-being and may indicate risk of depression.

SECONDARY OUTCOMES:
Polysomnography (PSG) for slow-wave sleep | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  PSG is an objective, overnight sleep study that records multiple physiological parameters to evaluate sleep architecture and detect sleep disorders. This study aims to use PSG to determine the amount of slow-wave sleep (SWS) among total sleep time. SWS, also known as deep sleep or NREM stage 3 (N3), is considered the most restorative stage of sleep. The normal range for SWS in adults is generally 10% to 20% of total sleep time, equating to about 40 to 110 minutes for those who sleep 7 to 9 hours per night.
Functional Magnetic Resonance Imaging (fMRI) | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  A non-invasive neuroimaging technique that measures brain activity by detecting blood oxygen level-dependent (BOLD) signal changes associated with neural activity. fMRI allows assessment of both task-related activation (e.g., responses to cognitive or emotional stimuli) and resting-state functional connectivity (e.g., interactions between large-scale brain networks). Key physiological indicators include:
  BOLD signal fluctuations reflecting regional brain activity. Functional connectivity metrics (e.g., correlations between brain regions). Task-related activation patterns in specific cortical and subcortical areas. Derived indices such as amplitude of low-frequency fluctuations (ALFF), regional homogeneity (ReHo), and network efficiency.
  Higher or more coherent activation/connectivity generally indicates more efficient neural processing, while abnormal patterns may suggest dysfunction in mood regulation, cognition, or sleep-wake processes.
non-invasive fiber optic physiological monitoring (nFOPT) for respiratory patterns | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  A novel non-invasive monitoring technique that uses fiber optic sensors to continuously measure physiological signals with high sensitivity and stability. This technology aims to investigate respiratory patterns during sleep. Higher irregularity in respiratory patterns may indicate poorer physiological regulation, while stable and coherent signals suggest healthier sleep and autonomic function.
Belun Ring for sleep apnea | The pretest will be conducted within one month prior to the intervention, and the posttest will be conducted within one month following the intervention.
  The prevalence and distribution of OSA across different severity levels will be evaluated using the apnea-hypopnea index/respiratory event index derived from the Belun Ring (bAHI). Belun Ring is a wearable, non-invasive device designed to continuously monitor physiological signals during daily life and sleep. It uses optical and motion sensors to provide detailed data on autonomic and sleep-related parameters. The severity of OSA is categorized based on the bAHI as follows: Normal: bAHI < 5 events/hour; Mild OSA: bAHI between 5 and 15 events/hour; Moderate OSA: bAHI between 15 and 30 events/hour; Severe OSA: bAHI > 30 events/hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol